CLINICAL TRIAL: NCT02721498
Title: Improving Outcome Measures For Physiotherapy Trials of Airway Clearance in Adults With Cystic Fibrosis
Brief Title: Improving Outcome Measures For Adult CF ACT Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2016CF001B
Record Dates: First submitted 2016-03-09; First posted 2016-03-29 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
Keywords: Respiratory Physiotherapy; Airway clearance techniques; Outcome measures
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visit A (Active Comparator): Rest period for 30-60 minutes
  Interventions: Other: Rest period
- Visit B (Active Comparator): Airway clearance session utilising the Active Cycle of Breathing techniques (ACBT) supervised by a specialist physiotherapist for 30-60 minutes.
  Interventions: Procedure: Airway clearance session using the Active Cycle of Breathing Techniques (ACBT)

INTERVENTIONS:
Procedure: Airway clearance session using the Active Cycle of Breathing Techniques (ACBT) — An airway clearance technique incorporating thoracic expansion exercises, breathing control (normal diaphragmatic breathing) and the forced expiration technique (or huffing)
  Arms: Visit B
Other: Rest period — A 30-60 minute of resting
  Arms: Visit A

SUMMARY:
This is a randomised controlled cross-over trial involving adult cystic fibrosis (CF) patients from the Royal Brompton Hospital, London investigating outcome measures used in airway clearance trials.

Each participant will attend the research facility for two visits. Participants will be randomly assigned to the order that they perform the study sessions. Visit A will involve a period of rest for up to 60 minutes in-between assessments; Visit B will involve a session of airway clearance (ACT) utilising ACBT supervised by a specialist physiotherapist in adult CF.

Participants will perform the outcome measure (OM) tests of impulse oscillation system (IOS), lung clearance index (LCI), and spirometry, then either rest (visit A) or perform a supervised ACBT session (visit B) using electronic impedance tomography (EIT) during the session. IOS, LCI and spirometry will be repeated after the session. Sputum will be collected throughout the ACT or rest sessions and for 30 minutes after each of these sessions is completed. Questionnaires asking patient views on the OMs will be completed at the end of each study visit.

Analysis will be based upon differences in outcome measures and in-between study days.

DETAILED DESCRIPTION:
Research Question: Does the use of a new assessment tool box (Electronic Impedance Tomography (EIT), Lung Clearance Index (LCI), Impulse Oscillation System (IOS)) give results that are more sensitive to change for the effect of an airway clearance technique (ACT) (the Active Cycle of Breathing Techniques (ACBT)) while having low variability and good repeatability in stable adult patients with cystic fibrosis (CF) than the traditional gold standard outcome measures of forced expiratory volume in one second (FEV1) and sputum wet weight?

Hypothesis: The use of a new outcome assessment tool box will allow more sensitive information about the effects of ACTs in stable adult patients with CF than the current gold standard measures.

This is a randomised controlled cross-over trial involving adult cystic fibrosis (CF) patients from the Royal Brompton Hospital, London. Participants will be their own controls. Each participant will attend the research facility for two visits. Prior to starting the study assessment session participants will be questioned to ensure they are in a stable state of their disease (characterised by symptoms and having had no treatment changes for 28 days prior to the visit). All participants will continue with the timing and prescribed dosing of all inhaled medications as directed prior to the study. Subjects will be their own controls. Subjects will be randomly assigned to the order that they perform the study sessions. Visit A will involve a period of rest for up to 60 minutes in-between assessments; Visit B will involve a session of airway clearance (ACT) utilising the Active Cycle of Breathing Techniques (ACBT) supervised by a specialist physiotherapist in adult CF. The ACT session will last for thirty minutes minimum, to 60 minutes maximum until a consensus is reached between participant and physiotherapist that the participant's chest is clear.

Subjects will perform the OM tests of impulse oscillation system (IOS), lung clearance index (LCI), and spirometry, then either rest (visit A) or perform a supervised ACBT session (visit B) using electronic impedance tomography (EIT) during the session. IOS, LCI and spirometry will be repeated immediately after the session. Sputum will be collected throughout the ACT or rest sessions and for 30 minutes after each of these sessions is completed. Questionnaires asking patient views on the OMs will be given for completion after the last OM test is completed on each study visit.

There are no planned follow up measurements for participants in this study design.

All usual medications will be permitted for this study. Attention will be paid to mucoactive drugs (Pulmozyme®, Mannitol®, Hypertonic saline) to ensure the same frequency and dosing of inhalations for both study visits.

Data will be analysed in 3 groups based upon disease severity. Analysis will be based upon differences in outcome measures and in-between study days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF (confirmed by standard criteria)
* Sixteen years of age or over
* Patients in a stable state (characterised by no required therapy changes within 28 days of visit and patient symptoms)

Exclusion Criteria:

* Current infective exacerbation or reduction in lung function requiring therapeutic intervention
* Current moderate haemoptysis (greater than streaking in the sputum)
* Current dependency on positive pressure support with ACT
* Previous history of spontaneous rib fractures
* Pregnancy
* Inability to give consent for treatment or measurement
* Current participation in another interventional study
* Current dependency upon non-invasive ventilation
* Current dependency upon oxygen therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in Lung Clearance Index | Immediately pre-intervention and immediately post-intervention
  This is a technique which involves breathing quietly through a tube whilst wearing nose clips. The test measures harmless tracer gases which are breathed in and out and measured by a sensitive gas-detection system. The LCI is calculated based on how long it takes for the gas to be breathed out from the lungs, and it shows if there are areas within the lung that are working less efficiently than others, for example when areas of the lung are clogged with mucus.
Change in Forced Expiratory Volume in One Second | Immediately pre-intervention and immediately post-intervention
  A forced expiratory manoeuvre into a spirometer (value derived from 1 second blow)
Electronic Impedance Tomography | During intervention
  This technique involves wearing a belt around the chest which has electrodes attached to it. Undetectable alternating electrical currents are then applied to the electrodes, which the participant will not be able to feel. The machine measures how easy or difficult it is for that current to travel through the lungs and any differences are calculated, giving a picture of the ventilation of the lung.
Change in Impulse Oscillation System | Immediately pre-intervention and immediately post-intervention
  The Impulse Oscillation system is a non-invasive technique where the participant breathes normally through a mouthpiece whilst wearing a nose clip, into a machine which produces small pressure vibrations (oscillations). The machine measures these vibrations and any changes to them to give an idea of obstructions to the airways, for example any mucus clogging.
Sputum Wet Weight | During intervention and for 30 minutes post-intervention
  Amount of sputum expectorated will be measured in a pre-weighed pot

SECONDARY OUTCOMES:
Change in Forced Vital Capacity | Immediately pre-intervention and immediately post-intervention
  A forced expiratory manoeuvre into a spirometer (value derived from full expiration)
Change in Forced Expiratory Flow at 25% of Forced Vital Capacity | Immediately pre-intervention and immediately post-intervention
  A forced expiratory manoeuvre into a spirometer (value derived from full expiration)
Change in Forced Expiratory Flow at 50% of Forced Vital Capacity | Immediately pre-intervention and immediately post-intervention
  A forced expiratory manoeuvre into a spirometer (value derived from full expiration)
Change in Forced Expiratory Flow at 75% of Forced Vital Capacity | Immediately pre-intervention and immediately post-intervention
  A forced expiratory manoeuvre into a spirometer (value derived from full expiration)
Oxygen saturation measurements | During interventions
  Completed via a finger probe connected to a pulse oximeter which will record saturations over the whole session.
Patient feedback questionnaire | Straight after the intervention
  A patient reported outcome investigating the opinions of participants on each of the OMs completed during the trial using open and Likert scale questions

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Simmonds, MD(Res) FRCP, Principal Investigator — The Royal Brompton & Harefield NHS Foundation Trust and Imperial College, London
Locations (1):
- The Royal Brompton Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kent L, Reix P, Innes JA, Zielen S, Le Bourgeois M, Braggion C, Lever S, Arets HG, Brownlee K, Bradley JM, Bayfield K, O'Neill K, Savi D, Bilton D, Lindblad A, Davies JC, Sermet I, De Boeck K; European Cystic Fibrosis Society Clinical Trial Network (ECFS-CTN) Standardisation Committee. Lung clearance index: evidence for use in clinical trials in cystic fibrosis. J Cyst Fibros. 2014 Mar;13(2):123-38. doi: 10.1016/j.jcf.2013.09.005. Epub 2013 Dec 5. PMID 24315208
- [Background] Bradley JM, Moran FM, Elborn JS. Evidence for physical therapies (airway clearance and physical training) in cystic fibrosis: an overview of five Cochrane systematic reviews. Respir Med. 2006 Feb;100(2):191-201. doi: 10.1016/j.rmed.2005.11.028. PMID 16412951
- [Background] Osman LP, Roughton M, Hodson ME, Pryor JA. Short-term comparative study of high frequency chest wall oscillation and European airway clearance techniques in patients with cystic fibrosis. Thorax. 2010 Mar;65(3):196-200. doi: 10.1136/thx.2008.111492. Epub 2009 Aug 23. PMID 19703826
- [Background] Pfleger A, Steinbacher M, Schwantzer G, Weinhandl E, Wagner M, Eber E. Short-term effects of physiotherapy on ventilation inhomogeneity in cystic fibrosis patients with a wide range of lung disease severity. J Cyst Fibros. 2015 Sep;14(5):627-31. doi: 10.1016/j.jcf.2014.12.017. Epub 2015 Jan 19. PMID 25612899
- [Background] Wettstein M, Radlinger L, Riedel T. Effect of different breathing aids on ventilation distribution in adults with cystic fibrosis. PLoS One. 2014 Sep 15;9(9):e106591. doi: 10.1371/journal.pone.0106591. eCollection 2014. PMID 25222606
- [Background] Horsley A. 2009. 'Non-Invasive Assessment of Ventilation Maldistribution in Lung Disease Using Multiple Breath Inert Gas Washouts', University of Edinburgh, UK
- [Background] Hurt, K. 2013. 'Small Airways Assessment In Adult Cystic Fibrosis', Imperial College (National Heart and Lung Institute), UK
- [Derived] Stanford G, Davies JC, Usmani O, Banya W, Charman S, Jones M, Simmonds NJ, Bilton D. Investigating outcome measures for assessing airway clearance techniques in adults with cystic fibrosis: protocol of a single-centre randomised controlled crossover trial. BMJ Open Respir Res. 2020 Oct;7(1):e000694. doi: 10.1136/bmjresp-2020-000694. PMID 33020113